CLINICAL TRIAL: NCT04921982
Title: The Efficacy of Traumatic Memory Modification Using a Memory Reconsolidation Procedure Under Propranolol Among Adolescents With Post-traumatic Stress Disorder
Brief Title: Efficacy of Traumatic Memory Modification Using Memory Reconsolidation and Propranolol Among Adolescents With PTSD
Acronym: PROPRADO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study could not begin within the period of validity of the authorizations. The project has been abandoned in its initially authorized form. The final study report will not be produced.
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35RC18_8852_PROPRADO
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Experimental)
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Oral administration of Propranolol, 90 minutes prior to a brief memory reactivation session, performed by a trained nurse once a week for six consecutive weeks.
  Arms: Propranolol
Drug: Placebo — Oral administration of Placebo, 90 minutes prior to a brief memory reactivation session, performed by a trained nurse, once a week for six consecutive weeks.
  Arms: Placebo

SUMMARY:
The aim of this study is to demonstrate the effectiveness of propranolol in blocking reconsolidation by reducing PTSD symptoms in the short and long term in adolescents with PTSD for more than 3 months.

ELIGIBILITY:
Inclusion Criteria:

* - Adolescents aged 12 to 18 years;
* Exposed to a single traumatic event or to events circumscribed in time, including sexual abuse in the absence of reminders in the environment;
* Fluent in French;
* Positive diagnosis of PTSD with the SCID-5;
* Disorders evolving for at least three months;
* Heart rate ≥ 55 bpm;
* Systolic blood pressure ≥ 100 mmHg;
* Written parental or legal guardian consent;
* Written agreement by the adolescent;
* Adolescents affiliated, via their parents, to the French social security body.

Exclusion Criteria:

* - Medical condition contraindicating administration of propranolol (COPD, asthma, cardio-vascular insufficiency, heart failure as second- and third-degree atrioventricular blocks, Prinzmetal angor, pheochromocytoma, Raynaud disease, history of an anaphylactic reaction, sinus node disease, hypoglycemia, AV blocks)
* Known chronic renal or hepatic insufficiency
* Schizophrenia;
* Mental retardation;
* Autism spectrum disorder;
* Acute severe suicidal ideation
* Traumatic brain injury (loss of consciousness > 10 minutes);
* Currently treated for substance or alcohol dependence;
* Currently treated for Attention Deficit Hyperactivity Disorder;
* Currently treated with a drug that can interfere with propranolol and that can represent a danger according to medical advice if it's suspended more than 24 hours.
* Currently treated with a bradycardic drug;
* Concurrent psychotropic medication with the exception of cyamemazine (suspended 48 hours before session)
* Concurrent trauma-focused psychotherapy in progress or stopped less than 1 month ago;
* Pregnancy or breast feeding.
* Current use of "recreative" toxic drugs
* Concurrent participation to another interventional study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change on score of PCL-5 | 7 weeks
  Difference on score on the PTSD Checklist for DSM-5 (PCL-5) between inclusion and one week after the end of treatment. PCL-5 is a 20-item self-report measure of the DSM-5 symptoms of PTSD used as a continuous measure. A decrease of 10 points on the PCL is usually considered as a clinically significant improvement. It has been used worldwide and among adolescents (Wang, 2015; Cao, 2017)

SECONDARY OUTCOMES:
Change on score of PCL-5 after each treatment session | 6 weeks
  Difference on score on the post-traumatic stress disorder Checklist for DSM-5 (PCL-5) between inclusion and after each dispensation of treatment. PCL-5 is a 20-item self-report measure of the DSM-5 symptoms of PTSD used as a continuous measure. A decrease of 10 points on the PCL is usually considered as a clinically significant improvement. It has been used worldwide and among adolescents (Wang, 2015; Cao, 2017) Scores consist of a total symptom severity score (from 0 to 80)
  Consistent with the likert scale:
  0 = Not at all
  1. = A little bit
  2. = Moderately
  3. = Quite a bit
  4. = Extremely Higher scores mean a worse outcome.
Change on score of PCL-5 at 3 months | 3 months
  Difference on score on the Post Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) between inclusion and 3 months after the beginning of the treatment. PCL-5 is a 20-item self-report measure of the DSM-5 symptoms of PTSD used as a continuous measure. A decrease of 10 points on the PCL is usually considered as a clinically significant improvement. It has been used worldwide and among adolescents (Wang, 2015; Cao, 2017) Scores consist of a total symptom severity score (from 0 to 80)
  Consistent with the likert scale:
  0 = Not at all
  1. = A little bit
  2. = Moderately
  3. = Quite a bit
  4. = Extremely
  Higher scores mean a worse outcome.
Change on score of PCL-5 at 6 months | 6 months
  Difference on score on the Post Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) between inclusion and 6 months after the beginning of the treatment. PCL-5 is a 20-item self-report measure of the DSM-5 symptoms of PTSD used as a continuous measure. A decrease of 10 points on the PCL is usually considered as a clinically significant improvement. It has been used worldwide and among adolescents (Wang, 2015; Cao, 2017) Scores consist of a total symptom severity score (from 0 to 80)
  Consistent with the likert scale:
  0 = Not at all
  1. = A little bit
  2. = Moderately
  3. = Quite a bit
  4. = Extremely
  Higher scores mean a worse outcome.
Change on score of PCL-5 at 12 months | 12 months
  Difference on score on the Post Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) between inclusion and 12 months after the beginning of the treatment. PCL-5 is a 20-item self-report measure of the DSM-5 symptoms of PTSD used as a continuous measure. A decrease of 10 points on the PCL is usually considered as a clinically significant improvement. It has been used worldwide and among adolescents (Wang, 2015; Cao, 2017) Scores consist of a total symptom severity score (from 0 to 80)
  Consistent with the likert scale:
  0 = Not at all
  1. = A little bit
  2. = Moderately
  3. = Quite a bit
  4. = Extremely Higher scores mean a worse outcome.
Change in CPC-DSM5 questionnaire score | 12 months
  Difference in functional impairment score of CPC-DSM5 at inclusion visit, before each dispensation of treatment (once per week for 6 weeks), one week after the end of treatment and 3, 6 and 12 months after the beginning of treatment. Functional impairment score will be assessed using CHILD PTSD CHECKLIST PARENT questionnaire. CPC is a self-questionnaire of 12 items. The total severity score ranges from 0 to 80 and is calculated by summing the ratings of the first 20 items. The CPSS-5-I also yields subscale scores for intrusion (Items 1-5), avoidance (Items 6-7), changes in cognition and mood (Items 8-14), and increased arousal and reactivity (Items 15-20).
  The interviewer rates the seven impairment items on a scale of 0 (not at all) to 4 (6 or more times a week/almost always), resulting in an impairment score that ranges from 0 to 28. The total impairment score does not contribute to the overall severity score.
Change in SCID-5 questionnaire score | 12 months
  Difference in Categorical diagnosis of PTSD using SCID-5 questionnaire at inclusion visit, before each dispensation of treatment (once per week for 6 weeks), one week after the end of treatment and 3, 6 and 12 months after the beginning of treatment. SCID-5 is for Structured Clinical Interview for DSM-5 is a semi-structured interview guide for making the major DSM-5 diagnoses used for the diagnosis of PTSD and depression.
Change in Child Depression Inventory score | 12 months
  Difference in Child Depression Inventory (CDI) score between inclusion visit and one week after the end of treatment, 6 months and 12 months after the beginning of treatment. There are 27 items quantifying symptoms such as depressed mood, hedonic capacity, vegetative functions, self-evaluation, and interpersonal behaviors. Each item consists of three statements graded in order of increasing severity from 0 to 2; children and adolescents select the one that characterized their symptoms best during the past 2 weeks. The item scores are combined into a total depression score, which ranges from 0 to 54. A higher CDI score means a higher depressive state.
Change in Adolescent Dissociative Experience scale | 12 months
  Difference in Adolescent Dissociative Experience (DES-A) score at inclusion visit, one week after the end of treatment, 6 and 12 months after the beginning of treatment. DES-A is a 28-items selfquestionnaire. Each item reaches to 0 (never happening) to 10 (always happening)
Change in Youth Self Report score | 12 months
  Scores for Behavioral and Somatic Disorders and for School/social functioning using Youth Self report (CBCL/YSR, parents/children) at inclusion visit , one week after the end of treatment, 6 and 12 months after the beginning of treatment. The YSR is a 112-item self-report designed for children and adolescents (ages 11-17) and largely used worldwide. It assesses behavioral competency and behavioral problems and parallels the Child Behavior Checklist (CBCL). The questionnaire provides scores for the following syndrome scales: anxious/depressed, withdrawn/depressed, somatic complains, social problems, thought problems, rule-breaking behavior, and aggressive behavior. The questionnaire provides scores for DSM-oriented scales.
  The YSR consists of 112 questions, scored on a three-point Likert scale (0=absent,
  1= occurs sometimes, 2=occurs often) Higher scores mean a worse outcome.
Change in suicidal riskk using Mini-Kid questionnaire | 12 months
  Difference in acute suicidal risk using Mini Kid questionnaire at inclusion visit , one week after the end of treatment, 6 and 12 months after the beginning of treatment. The Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI Kid) is a short, structured diagnostic interview for DSM-IV and ICD-10 psychiatric disorders in children and adolescents. Only part C will be used to assess diagnosis of acute suicidal risk. Scores reaches from 0 to 10 Higher scores mean a worse outcome.
Evaluation of the tolerance to treatment | 6 weeks
  Evaluation of the tolerance to treatment at each dispensation of treatment (once per week for 6 weeks) by the research nurse: Clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Dayan, Pr, Principal Investigator — CHU Rennes
Locations (10):
- France (10):
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CH Bohars, Bohars
  - AP-HP Louis Mourier, Colombes
  - CH Le Havre, Le Havre
  - CHU Limoges, Limoges
  - CHU Nantes, Nantes
  - CHU Poitiers, Poitiers
  - CH Guillaume Régnier, Rennes
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No